CLINICAL TRIAL: NCT00752843
Title: A Phase I, Open-Label, Fixed-Sequence Study to Determine the Effect of Single and Multiple Oral Doses of CORLUX (TM) (Mifepristone) on the Pharmacokinetics of a Single Oral Dose of Fluvastatin (a CYP2C9 Probe) in Healthy Volunteers
Brief Title: A Phase I Study to Determine the Effect of Mifepristone on the Pharmacokinetics of Fluvastatin in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Corcept Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: C-1073-16
Record Dates: First submitted 2008-09-12; First posted 2008-09-16 (Estimated); Last update posted 2012-02-17 (Estimated); Status verified 2012-02

CONDITIONS: Healthy Subjects
Keywords: mifepristone; CORLUX; fluvastatin; Lescol; drug-drug interaction; DDI; pharmacokinetics
MeSH Terms: interventions — Mifepristone; Fluvastatin; Corlux

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: mifepristone + fluvastatin

INTERVENTIONS:
Drug: mifepristone + fluvastatin — Subjects will receive a single oral dose of 40 mg PO of fluvastatin on three occasions: alone (Day 1), at the same time as a single dose of CORLUX 1200 mg (Day 8) and during concomitant administration of CORLUX 1200 mg/day (CORLUX on Days 8-14, fluvastatin on Day 14).
  Other Names: CORLUX + Lescol

SUMMARY:
This study is to determine the effect of single and multiple oral doses of mifepristone on the pharmacokinetics of a single oral dose of fluvastatin administered to healthy volunteers.

DETAILED DESCRIPTION:
This is a fixed-sequence, drug-drug interaction study in healthy volunteers lasting up to a total of 9 weeks: up to 4 weeks screening, approximately 2 weeks for dosing (including a 1-week washout between periods), and approximately 3 weeks of a drug-free interval until termination. The purpose of this study is to determine the effect of single and multiple oral doses of CORLUX on the pharmacokinetics of a single oral dose of fluvastatin administered to healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Male or female healthy volunteers
* Body mass index (BMI) of 18-32 kg/m2
* Female subjects must have a negative serum pregnancy test result prior to entry into the study
* All female subjects must not be of child-bearing potential
* All male subjects with female partners of childbearing potential must consent to use a medically acceptable double-barrier method of contraception and not donate sperm throughout the study period and for at least 3 months (90 days) after the last dose of study medication
* The subject agrees to abstain from grapefruit or grapefruit juice for at least 2 weeks prior to the first dose and until completion of the pharmacokinetic sampling (Day 15)
* The subject must be able to provide written informed consent

Exclusion Criteria:

* Any acute or chronic disease state, including but not limited to cardiovascular, dermatological, endocrine, gastrointestinal, hepatic, pulmonary, and renal conditions determined to be clinically significant by the Investigator
* Any clinically significant abnormal clinical laboratory tests as determined by the Investigator
* Any concomitant medications (including prescription, over-the-counter or illicit) within either 30 days or five half-lives (whichever is shorter) prior to dosing
* Positive urine drug screen for any illicit drugs
* Use of tobacco or any nicotine-containing products during the previous three months
* Grapefruit juice within two weeks prior to first dose
* Participation in a clinical investigation of any drug, biological or other investigational therapy within 30 days prior to dosing
* Signs and/or symptoms such as orthostatic hypotension, fatigue, anorexia, nausea, abdominal pain, joint and muscle pain if considered to be a marker of adrenal insufficiency
* History of an allergic reaction to mifepristone or fluvastatin
* Positive serum test for human immunodeficiency virus (HIV), hepatitis B virus or hepatitis C virus
* Blood donation within 30 days of dosing

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-09; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
To determine the effect of single and multiple oral doses of CORLUX on the pharmacokinetics of a single oral dose of fluvastatin administered to healthy volunteers. | 8, 9, 12, 13, 14, & 15 days

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Swearingen, MD, Principal Investigator — MDS Pharma; Thaddeus Block, MD, Study Director — Corcept Therapeutics
Locations (1):
- MDS Pharma, Tempe, Arizona, United States

REFERENCES:
- See also: Corcept Therapeutics — http://www.corcept.com
- See also: MDS Pharma — http://www.mdsps.com